CLINICAL TRIAL: NCT03343327
Title: A Single Centre, Open-label, Randomised, Single Dose, Two Period, Crossover Relative Bioavailability Study of Chronocort® Versus Cortef® Immediate Release Hydrocortisone Tablets in Dexamethasone-suppressed Healthy Adult Male Subjects.
Brief Title: A Study of Chronocort® Versus Cortef ® in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry); Brush Clinical Research Ltd. (Industry); Voet Consulting (Industry); Bionical Emas Ltd. (Unknown); Medical Matters International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-008
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chronocort®, then Cortef® (Experimental): Single dose of 20mg Chronocort® (oral administration), followed by a single dose of 20mg Cortef® Immediate Release Hydrocortisone Tablets (oral administration).
  Interventions: Drug: Chronocort®; Drug: Cortef®
- Cortef®, then Chronocort® (Active Comparator): Single dose of 20mg Cortef® Immediate Release Hydrocortisone Tablets (oral administration), followed by a single dose of 20mg Chronocort® (oral administration).
  Interventions: Drug: Chronocort®; Drug: Cortef®

INTERVENTIONS:
Drug: Chronocort® — Single dose of 20mg Chronocort® administered in one treatment period
Drug: Cortef® — Single dose of 20mg Cortef® administered in one treatment period

SUMMARY:
This was a single centre, open label, randomised, two period, crossover study to evaluate the bioavailability of Chronocort® versus Cortef® immediate release hydrocortisone tablets in dexamethasone-suppressed healthy adult male subjects.

DETAILED DESCRIPTION:
This study was an open-label, randomised, single dose, two-period, crossover study in 25 healthy male subjects.

The study comprised of a pre-study screen, followed by 2 treatment periods (1 and 2) and a post-study followup.

Screening (Day -28 to Day -1): Screening assessments were carried out within 28 days before first administration of IMP. Eligible subjects were asked to return for the treatment periods. Continued eligibility was confirmed pre-dose during each treatment period.

Treatment Periods (Day -1 to Day 1): Eligible subjects received a single-dose of each IMP over 2 treatment periods (1/period as determined by the randomisation schedule), each separated by 7 days washout. Each study period was approximately 2 days in duration, from the afternoon of Day -1 to the morning of Day 1 at 24 hours (h) post-dose. During each treatment period, Subjects arrived at the Clinical Unit on Day -1, IMP was administered on the morning of Day 0 fasted (following an overnight fast of at least 10 h) and subjects were discharged following the 24 h post-dose blood samples and completion of the scheduled measurements.

Pharmacokinetic (PK) samples were collected pre-dose at ~ -2min and up to 23 h post-dose (Day 1) (24 samples) for the measurement of cortisol. A further 3 baseline samples were taken for the measurement of cortisol. Safety was also evaluated throughout the study.

Post Study: After completion of both study periods, the subjects returned 4-22 days later for the final followup visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 45 years of age inclusive (at screening).
2. A BMI of 18-30 kg/m2 (inclusive).
3. No clinically significant abnormal serum biochemistry, haematology or urine examination values as defined by the Investigator.
4. A negative urinary drugs of abuse screen. A positive alcohol test or drugs of abuse test may be repeated at the discretion of the Investigator.
5. Negative HIV and Hepatitis Band C results.
6. No clinically significant abnormalities in 12-lead ECG as defined by the Investigator.
7. No clinically significant deviation outside the normal ranges for blood pressure and heart rate measurements as defined by the Investigator.
8. Subjects (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) and sexual partners must use 2 effective contraception methods during the trial and for 3 months after the last dose, for example:

   * Oral, injected or implanted hormonal contraceptive+ condom
   * Intra-uterine device (IUD) + condom
   * Diaphragm with spermicide + condom
9. Subjects must be available to complete both periods of the study and the follow-up visit.
10. Subjects must satisfy a medical examiner about their fitness to participate in the study.
11. Subjects must be able to read and understand the informed consent form and must provide written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Receipt of any medication with the exception of paracetamol within the 14 days prior to dosing (including topical steroids, vitamins, dietary supplements or herbal remedies).
3. Evidence of renal. hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. Receipt of any vaccination within the previous one month.
5. Presence of infections (systemic fungal and viral infections, acute bacterial infections).
6. Current or previous history of tuberculosis.
7. A clinically significant history of previous allergy/sensitivity to hydrocortisone and/or dexamethasone.
8. Meeting any of the contraindications for Cortef® and/or dexamethasone, as detailed in the United States Prescribing Information (USPI)/Summary of Product Characteristics (SmPC), respectively
9. A clinically significant history of drug or alcohol abuse.
10. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
11. Participation in a New Chemical Entity clinical study or a marketed drug clinical study within the previous three months, or five half- lives of the study drug, whichever is the longer period. (NB. the three-month washout period between trials is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
12. Subjects who have consumed more than two units of alcohol per day within seven days prior to the first dose or have consumed any alcohol within the 48-hour period prior to the first dose.
13. Donation or receipt of 450 mL of blood within the previous three months.
14. Subjects who smoke (or ex-smokers who have smoked within six months prior to first dose). This includes e-cigarette and shisha users.
15. Subjects who work shifts (i.e. regularly alternate between days, afternoons and nights).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve from time 0 to infinity (AUC0-inf) of Chronocort® to Cortef® based on baseline adjusted and unadjusted serum cortisol concentration calculated for each sampling time point. | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  Comparing the area under the concentration time curve of Chronocort® compared to Cortef® immediate release hydrocortisone tablets.

SECONDARY OUTCOMES:
Pharmacokinetic parameters for serum cortisol + relative bioavailability - Cmax | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  The following PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
  ◦ Cmax Maximum plasma cortisol concentration.
Pharmacokinetic parameters for serum cortisol + relative bioavailability - Tmax | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  The following PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
  ◦ Tmax The time to maximum observed cortisol concentration sampled during a dosing interval.
Pharmacokinetic parameters for serum cortisol + relative bioavailability - Kel | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  The following PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
  ◦ kel Elimination rate constant.
Pharmacokinetic parameters for serum cortisol + relative bioavailability - t1/2 | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  The following PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
  ◦ t1/2 Terminal half-life.
Pharmacokinetic parameters for serum cortisol + relative bioavailability - AUC0-t | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  The following PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
  ◦ AUC0-t Area under the plasma cortisol concentration-time curve (AUC) from the time of dosing to the time of the last observed concentration.
Pharmacokinetic parameters for serum cortisol - Serum cortisol clearance (CL/F) | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  Calculated as Dose / AUC0-inf. This PK endpoint was derived from baseline adjusted and unadjusted serum cortisol concentration-time data following administration of each IMP.
Pharmacokinetic parameters for serum cortisol - Distribution during terminal elimination (Vz/F) | Samples taken at 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 11,12, 13, 14, 16, 18, 20, 22, and 24 hours (morning of Day 1) in both periods.
  Volume of distribution based on the terminal elimination phase following extravascular administration derived from baseline adjusted and unadjusted serum cortisol
Observed changes in Safety Laboratory Data | Screening, Pre-dose and 10h and 24h post-dose during both treatment periods; Follow up
  Observed changes in Safety Laboratory data (biochemistry, haematology & urinalysis) during the course of the study, with any out of normal range values flagged.
Observed changes in Vital Signs | Screening; Pre-dose and at 4 and 10h post-dose during both treatment periods; Follow up
  Observed changes in vital signs data (blood pressure, pulse rate and oral temperature) during the course of the study, with any out of normal range values flagged.
Observed changes in Electrocardiogram (ECG) data during the course of the study | Screening, Pre-dose and 10h post-dose during both treatment periods; Follow up
  12-Lead ECG parameters (Heart Rate, PR interval, QRS width, QT interval, and QT interval corrected using Bazett's formula (QTcB)) and investigator clinical interpretation was listed with any out of normal range values flagged.
Adverse Events | Through study completion - approximately 6 weeks
  Adverse events (AEs) observed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: A Koch, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd., Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No